CLINICAL TRIAL: NCT00834457
Title: A Pilot Study Of the Effects of Highly Active Antiretroviral Therapy on Kaposi's Sarcoma in Zimbabwe
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Parirenyatwa Hospital (Other)
Collaborators: University of Colorado, Denver (Other); GlaxoSmithKline (Industry); Abbott (Industry)
Responsible Party: Principal Investigator, Margaret Borok, Principal Investigator, Parirenyatwa Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COL30512
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: AIDS-related Kaposi's Sarcoma
Keywords: AIDS-related Kaposi's sarcoma; antiretroviral therapy
MeSH Terms: conditions — AIDS-related Kaposi sarcoma | interventions — abacavir, lamivudine, and zidovudine drug combination; abacavir; abacavir, lamivudine drug combination; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2A (Active Comparator): co-formulated abacavir 300mg/3TC 150mg/zidovudine 300mg po(Trizivir)one tablet twice daily(BID)for 96 weeks
  Interventions: Drug: abacavir/3TC/zidovudine
- 2B (Active Comparator): co-formulated abacavir 600mg/3TC 300mg orally (as Kivexa) one tablet daily plus fixed dose lopinavir 133.3mg/ritonavir 33.3mg orally (as Aluvia) four tablets daily for 96 weeks
  Interventions: Drug: abacavir /3TC plus ritonavir boosted lopinavir

INTERVENTIONS:
Drug: abacavir/3TC/zidovudine — continued use of oral co-formulated abacavir 300mg/3TC 150mg/zidovudine 300mg for 96 weeks
  Other Names: Trizivir
  Arms: 2A
Drug: abacavir /3TC plus ritonavir boosted lopinavir — fixed dose abacavir 600mg/3TC 300mg one tablet po QD for 96 weeks plus fixed dose ritonavir 33.3mg/lopinavir 133.3mg four tablets po QD for 96 weeks
  Other Names: Kivexa or Epzicom; Aluvia
  Arms: 2B

SUMMARY:
Open-label study of a regimen of antiretrovirals for the treatment of AIDS-KS. This study will be conducted at a single site, the Parirenyatwa Hospital KS Clinic.

Step 1 was conducted to determine the extent of clinical resolution of AIDS-KS disease in response to treatment with antiretroviral therapy and to investigate whether clinical resolution of KS is associated with suppression of KSHV replication.

Step 2 was developed to then evaluate the clinical, immunological, and virological effects of a switch from a twice-daily all-nucleoside reverse transcriptase inhibitor (NRTI) antiretroviral regimen to a once-daily regimen of 2 NRTIs plus a ritonavir-boosted protease inhibitor in persons with AIDS-KS and good virologic suppression an all NRTI regimen.

Step 3 was included to evaluate the clinical, immunological, and virological effects of intensification with a ritonavir-boosted protease inhibitor in persons with AIDS-KS who have virological failure on an all NRTI regimen.

DETAILED DESCRIPTION:
To identify factors associated with successful treatment of KS with antiretroviral therapy and to determine if highly active antiretroviral therapy improves survival and quality of life for persons with AIDS-KS in Zimbabwe.

A secondary objective is to investigate the durability of HIV-1 suppression by the combination of ABC/3TC/ZDV in persons infected with HIV-1 subtype C and to evaluate the timing and characteristics of mutations in HIV-1 reverse transcriptase in subjects who fail to achieve, or to maintain suppression of HIV-1 replication during treatment with ABC/3TC/ZDV.

An important objective is to assess adherence to a simplified antiretroviral regimen in a resource-limited setting.

The study will evaluate the clinical, immunological, and virological effects of a switch from a twice-daily all-nucleoside reverse transcriptase inhibitor (NRTI) antiretroviral regimen to a once-daily regimen of 2 NRTIs plus a ritonavir-boosted protease inhibitor in persons with AIDS-KS and good virologic suppression on ABC/3TC/ZDV (see above).

ELIGIBILITY:
Inclusion Criteria:Completion of at least 96 weeks of treatment with ABC/3TC/ZDV on protocol Step 1.

* Currently receiving ABC/3TC/ZDV on Step 1/initial open-label allNRTI phase of study.
* Plasma HIV-1 RNA < 400 copies/mL on the most recent plasma HIV-1 RNA performed within 4 weeks of Step 2 entry.
* Willing to potentially switch to a new antiretroviral regimen.
* In the opinion of the site investigator currently has clinical evidence of active KS disease.

Exclusion Criteria

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Compare effects of twice-daily all-(NRTI) antiretroviral regimen to a once-daily regimen of 2 NRTIs plus a protease inhibitor AIDS-KS subjects with good virologic suppression on all-NRTI regimen. | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Z Borok, FRCP, Principal Investigator — University of Zimbabwe College of Health Sciences Department of Medicine; Thomas B Campbell, MD, Study Chair — University of Colorado, Denver
Locations (1):
- University of Zimbabwe College of Health Sciences Department of Medicine, Harare, Zimbabwe